CLINICAL TRIAL: NCT02958072
Title: LeucoPatch in Malleoli Ulcer Study
Acronym: LiDMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Reapplix (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LiDMUS
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Malleoli Ulcers; Malleoli Ulcers
Keywords: Malleoli ulcers; Diabetes; Healing; Dressing; LeucoPatch
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- LeucoPatch (Experimental): Treatment with usual ulcer care and LeucoPatch once weekly up til 24 weeks or until healing.
  Interventions: Other: LeucoPatch
- Usual care followed by LeucoPatch (Active Comparator): Usual care weekly for 12 weeks, if the ulcer persist after the12 weeks LeucoPatch treatment will be started for up to 12 weeks or until healing.
  Interventions: Other: LeucoPatch

INTERVENTIONS:
Other: LeucoPatch — LeucoPatch is an fully autologous growth factor-containing dressing

SUMMARY:
An International Multicenter study evaluation, off the effect of the fully autologous growth factor-containing patch LeucoPatch, on healing of recalcitrant malleoli ulcers.

To compare the impact of LeucoPatch as part of usual care in multidisciplinary Foot clinic settings, versus usual care in the same clinics on malleoli ulcers healing.

DETAILED DESCRIPTION:
Diabetic Foot Ulcers are a common and severe complication, that affects Patients Life Quality. Healing time is often long and the Diabetic foot ulcer is the dominating not traumatic reason for leg amputation.

Treatment of a diabetic foot ulcer requires debridement, offloading, regularly foot care, specially tailored shoes, antimicrobial treatment, and sometimes even surgical interventions. Despite all these interventions the diabetic foot ulcer may not heal.

Malleoli ulcers in patients without diabetes share several features of pathogenesis and lack of healing potentials with the Diabetic Ulcer. Like the features of pathogenesis and lack of healing potential and are therefore included in this study.

Research has shown that other methods such as Growth factors may be a way to enhance the chance of healing.

Growth Factors have been shown to have a positive effect in studies, but no products that are characterized as autologous have as yet obtained positive results in controlled studies.

LeucoPatch is produced solely from a patient´s own blood without addition, and is autologous. LeucoPatch appears as an elastic membrane and can be fitted to the individual ulcer.

LeucoPatch is shown to contain as many or more growth factors as existing products, and has a high concentration of fibrin, platelets and leukocytes.

A non-controlled study was made on ulcers less than 10cm 2 and 52% had competed epithelization after 20 weeks. An International randomized multicenter trial is ongoing to evaluate the efficacy and safety of LeucoPatch on healing of hard to heal diabetic foot ulcers below the malleoli.

This Study is designed to test the healing effect of the LeucoPatch on malleoli ulcers, the Patient will be randomized and the healing will be confirmed by a blinded observer.

ELIGIBILITY:
Inclusion Criteria:

* Foot ulcer at the malleoli area between 0,25 cm² and 5,0 cm²
* Foot ulcer duration more than 6 weeks
* No need for arterial revascularisation- as judged by the Investigator
* informed consent

Exclusion Criteria:

* Hemoglobin concentration under 6.5 mmol/l screening
* Non-compliant with blood-letting
* Clinically infected ulcer
* Patient planned for or has had a revascularization procedure in the affected leg within the last 8 weeks
* The ulcer have been treated with growth factors in the last 8 weeks
* History of deep venous insufficiency, chronic venous leg ulcer or stasis dermatitis
* Breast-feeding women or fertile women not agreeing to use an effective method of contraception
* Participation in another clinical ulcer-healing study within the last 4 weeks
* Patient has previously been randomized in this study
* Judgement by the investigator that the patient is not able to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2023-03 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Healing of malleoli ulcer (YES/NO) | up to 24 weeks of treatment
  Confirmed by a blinded observer

SECONDARY OUTCOMES:
Time to healing of malleoli ulcer | 24 weeks
  Weeks from Inclusion to Wound healing
Ulcer area reduction based on Image J measured on acetate drawing | 24 weeks
Health related quality of life questionnaire SF12 | week 0, week 12, and week 24
  Short Form 12 questionnaire (quality of life)SF-12
Health related quality of life questionnaire EQ-5D | week 0, week 12, and week 24
  Euroquol-D5 questionnaire(mood and function) EQ-5D
Pain at ulcer location | week 0, week 6, week 12 and week 24
  VAS Score (Visual Analogue Scale)
Z scores of combined plasma concentration of growth factors, cytokines and inflammatory markers | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lise Tarnow, Professsor, Study Director — Nordsjaellands Hospital
Locations (6):
- Denmark (5):
  - Bispebjerg hospital, Copenhagen, Capital Region
  - Viborg Sygehus, Viborg, Region Midt
  - Nordsjaellands Hospital, Hillerød, Regionh
  - Herlev-Gentofte Hospital, Herlev
  - Kolding Sygehus, Kolding
- Skaane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No